CLINICAL TRIAL: NCT00758823
Title: Randomized Controlled Trial Comparing Efficacy and Tolerance of Four Pediculicides Acting Mechanically With Reference Product Acting Chemically (Prioderm)
Brief Title: Randomized Controlled Trial Comparing Efficacy and Tolerance of Four Pediculicides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omega Pharma (Industry)
Responsible Party: Maureen Tytgat/Plant Manager, Omega Pharma
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: OMEGA-IZ2008-V6
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Headlice Infections
Keywords: head lice

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Paranix — pediculicide product
  Other Names: Paranix Spray; Paranix Mousse; Paranix Lotion; Hedrin

SUMMARY:
THe main goal of our randomized controlled trial with blinded observer will be to compare four pediculicide products acting mechanically, Paranix Spray, Paranix Lotion, Paranix Mousse and Hedrin against a reference product acting chemically, Prioderm, during a non-inferiority (20% equivalence). THe randomization will be balanced every 10 families. The secondary objective will be to compare the lenticide efficacy of the products and their local tolerance and cosmetic acceptibility.

ELIGIBILITY:
Inclusion Criteria:

* Subject-male or female, child > 3 years and adult
* Pediculosis of scalp, confirmed by the identification of minimum 5 live lice with a fine-tooth comb
* Negative urine pregnancy test before inclusion for women of childbearing potential
* Use of a contraceptive method by hormonal contraceptives or IUDs or tubal ligation or condoms for women of childbearing potential
* Subject agreeing to participate in the study with written informed consent for participation
* Written consent of both parents for the minor patients.

Exclusion Criteria:

* Children under 3 years.
* Woman pregnant or lactating or without contraception
* Use of a pediculicide or lenticide treatment within 2 weeks before entry into the study
* Subject with known hypersensitivity to any component of the tested products
* Subject who participated in a clinical study in the 3 months prior to inclusion
* Ongoing treatment potentially interacting with the treatment under study (other pediculicide products)
* Subject undertreatment susceptible to influence the evaluation of the trial (including trimethoprim-sulfamethoxazole).
* Severe medical or psychiatric illness considered by the investigator as potentially dangerous to the subject or incompatible with the conduct of the study
* Asthma
* Subject unable for linguistic or psychiatric reasons to understand the information and give informed consent
* Subject refusing to give written consent
* Subject deprived of his liberty by administrative or judicial decision, or guardianship
* Patient hospitalized in a medical or social facility for another reason that biomedical research

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
statistical analysis will compare the number of successes and failures for each products | Day 1, Day 7 and day 14

CONTACTS AND LOCATIONS:
Overall Officials: Claire Bouges-Michel, MD, MCU-¨H, Principal Investigator — Parasitology-Mycology, APHP, CHU Avicienne; Rexline, Dr. Sr., Principal Investigator — St. Thomas Hospital
Locations (1):
- St. Thomas Hospital, Chennai, Tamil Nadu, India